CLINICAL TRIAL: NCT01475578
Title: A Randomized, Double-Blind, Double-Dummy, Active-Controlled, Parallel, Comparative, Multicenter, Phase II Study to Evaluate the Efficacy and Safety of STA-1 Capsule in Patients With Vascular Dementia (Marrow-Sea Deficiency)
Brief Title: Study of STA-1 Capsule in Patients With Vascular Dementia (Marrow-Sea Deficiency)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sinphar Pharmaceutical Co., Ltd (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2001ZL272
Record Dates: First submitted 2011-11-14; First posted 2011-11-21 (Estimated); Last update posted 2011-11-21 (Estimated); Status verified 2011-11

CONDITIONS: Vascular Dementia
Keywords: Vascular Dementia
MeSH Terms: conditions — Dementia, Vascular | interventions — Ergoloid Mesylates

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- STA-1 (Experimental): STA-1 capsule (Cistanche tubulosa), 2 capsules/time, 3 times/day, orally
  Dummy Ergoloid Mesylates tablet (Placebo), 2 tablets/time, 3 times/day, orally
  Interventions: Drug: STA-1
- Ergoloid Mesylates (Active Comparator): Ergoloid Mesylates tablet, 2 tablets/time, 3 times/day, orally before meal
  Dummy STA-1 capsule (Placebo), 2 capsules/time, 3 times/day, orally
  Interventions: Drug: Ergoloid Mesylates tablet

INTERVENTIONS:
Drug: STA-1 — STA-1 capsule (manufactured by Sinphar Tian-Li (Hangzhou) Pharm. Co., Ltd.; Batch number: 020121), 2 capsules/time, 3 times/day, orally
  Arms: STA-1
Drug: Ergoloid Mesylates tablet — Ergoloid Mesylates tablet (manufactured by Tianjin Huajin Pharmaceutical Factory; Batch number: 011230), 2 tablets/time, 3 times/day, orally before meal
  Arms: Ergoloid Mesylates

SUMMARY:
The objectives of this phase II study of STA-1 capsule was to make preliminary evaluation on clinical efficacy and safety of STA-1 capsule in order that based on the dosage and study structure planned in this project, the dosage and study structure of phase III study can be confirmed.

DETAILED DESCRIPTION:
This phase II clinical trial was planned to be in double-blind, double-dummy, active-controlled, parallel, comparative, multicenter design. Two hundred and 40 eligible subjects were planned to be recruited by 5 study centers. The treatment period planned in the protocol was 3 months with 5 study visits including Randomization visit (Day 0), three post-treatment visits (1 and 2 months after Randomization visit and Final visit) and 1 follow-up visit made at 6 month after Randomization visit.

After subjects recruited by this study having read and singed the ICF, they were arranged to be collected information of demographics, medical history, allergy history, medication history, and concomitant medication. Laboratory and physical examination including vital signs were performed, and Hachinski Ischemia Score (HIS), Mini-Mental Status Examination (MMSE), and Classification of Marrow-Sea deficiency were evaluated to ensure subject's eligibility to enter this study. After the subjects were confirmed eligible, they were randomly assigned to either STA-1 or Ergoloid Mesylates group. Blessed-Roth Behavior Scale (BBS) and Activities of Daily Living (ADL) Scale were measured after subjects were randomized. These subjects were then dispensed study medications for 1-month use.

The eligible subjects were requested to bring back unused study medication, if any, to study centers at 1, 2, and 3 months (Final visit) after the Randomization visit. At these visits, measurements of MMSE, BBS, ADL scales, and Classification of Marrow-Sea deficiency were collected. Information concomitant medications and AEs were also recorded. Physical and laboratory examinations were performed at Final visit. Each subject was dispensed with study medications for his/her subsequent treatment period at month-1 and -2 visits. Unused study medications were collected with drug accountability documented. Subjects were dismissed from the study at the Final visit.

Subjects were measured MMSE, BBS, and ADL scales at 6 months after the Randomization visit if they were available for follow-up evaluations.

ELIGIBILITY:
Inclusion Criteria:

1. Meeting criteria of dementia according to Diagnostic and Statistical Manual of Mental Disorders, fourth edition (DSM-IV)
2. Meeting criteria of vascular dementia according to National Institute of Neurological Disorders and Stroke-Association Internationale pour la Recherche et l'Enseignement en Neurosciences (NINDS/AIREN)
3. With Mini-Mental State Examination (MMSE score) ≦17 (illiteracy); ≦20 (elementary school); ≦24 (high school or above)
4. With Hachinski's ischemic score (HIS) ≧7
5. With marrow-sea deficiency from Chinese medicine's perspective
6. Classified mild to moderate dementia based on MMSE score
7. With body weight 45 to 95 Kg
8. Aged 45 to 80 years old (inclusive). Either gender is eligible. Female subjects must be postmenopausal (for at least 1 year) women without fertility
9. Having signed informed consent form
10. Correct understanding of pharmaceutical research and good compliance to study personnel's observation and evaluation

Exclusion Criteria:

1. Dementia besides study indication based on DSM-IV and NINDS/AIREN, e.g. Alzheimer's disease, Lwey body disease, etc.
2. With HIS < 7
3. Diagnosed significant depression based on DSM-IV with score >8 or with other mental diseases/disorders
4. With cognitive dysfunction caused by head impairment
5. With medical history of epilepsy, encephalitis, or any other diseases that may result in dementia, e.g. Parkinson's disease, Huntington disease, Pick disease, etc. Patients with epilepsy attacked occasionally should be examined at the first visit by electroencephalography (EEG) and should be excluded from this study if by the test results are positive.
6. With certain diseases that may interfere the evaluation of cognitive function, including abuse of alcohol, or DSM-IV diagnosed abuse of drugs or mental drugs in past 5 years. Severe anemia patients should also be excluded.
7. With severe mental dysfunction, e.g. hemiplegia, aphasia, visually and hearing impairment, etc.
8. With cardiac disorder, e.g. heart rate ≦ 50 or ≧ 180 times/minute
9. With supine or sitting Systolic blood pressure ≦ 100 or ≧ 180 mmHg
10. With other disease, especially hepatic, renal, or cardiac disorders, e.g. ALT/SGPT or AST/SGOT > 3 times of upper limit of normal range, serum creatinine > 177 umol/L (2mg/dL), or congestive heart failure (cardiac function 2-4 in classification)
11. With malignant neoplasm
12. With thyroid dysfunction or syphilis
13. Failed to control diabetes. Diabetes patients can not enter the study unless the status becomes stable through dietary modification, taking hypoglycemic agents, or receiving insulin.
14. With asthma or chronic obstructive pulmonary disease
15. With multiple neuritis
16. With myasthenia gravis and amyotrophic
17. With severe indigestion, or gastrointestinal obstruction, or gastric and duodenal ulcer, or other gastrointestinal diseases that can affect drug absorption
18. With glaucoma
19. Ever attending other clinical trials in past 30 days

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2002-03; Primary Completion 2002-10 (Actual); Study Completion 2002-10 (Actual)

PRIMARY OUTCOMES:
Changes from Baseline in Mini-Mental State Examination (MMSE) | Month 1, Month 2, , Month 3, , Month 6
  MMSE were used to evaluate subject's change in orientation, attention and calculation, immediate recall and delayed memory, and language ability before and after treatment.
Changes from Baseline in Blessed-Roth Behavior Scale (BBS) | Month 1, Month 2, , Month 3, , Month 6
Changes from Baseline in Activities of Daily Living (ADL) | Month 1, Month 2, , Month 3, , Month 6

SECONDARY OUTCOMES:
Changes from Baseline in the symptom scales from Chinese medicine's perspective | Month 1, Month 2, , Month 3, , Month 6

CONTACTS AND LOCATIONS:
Overall Officials: Mingjun Yang, Study Chair — Affiliated Hospital of Chengdu University of Traditional Chinese Medicines
Locations (5):
- China (5):
  - Affiliated Hospital of Chengdu University of Traditional Chinese Medicines, China, Chengdu
  - Fujian Academy of Traditional Chinese Medicine, Fujian
  - Hospital (Traditional Chinese Medicine) Affiliated to Luzhou Medical College, Luzhou
  - Affiliated Hospital of Shaanxi Academy of Traditional Chinese Medicine,, Shaanxi
  - Xi'an Traditional Chinese Medicine Hospital, Xi'an